CLINICAL TRIAL: NCT02137980
Title: Registry of Non-primary Angioplasty at Hospitals Without Surgery On-site
Acronym: CPORT
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: NA_00046362
Record Dates: First submitted 2014-03-18; First posted 2014-05-14 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Coronary Artery Disease; Heart Attack; Angina
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction; Angina Pectoris

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a simple registry of patients undergoing PCI at hospitals without surgery on-site who were participants in the CPORT-E project. The aim of the registry is simple data collection and reporting to respective State Departments of Health. The registry population consists of patients undergoing diagnostic cardiac catheterization for suspected CAD at hospitals without SOS and who require PCI.

ELIGIBILITY:
Inclusion Criteria:

Patient inclusion criteria are:

Pre-catheterization

1. must be undergoing diagnostic cardiac catheterization for suspected CAD
2. be at least 18 years of age
3. must not be pregnant (negative pregnancy test) or must not be of childbearing potential
4. must be able to give informed consent. Post-catheterization
5. coronary artery disease judged to be clinically and angiographically significant
6. ability to perform PCI with equipment available at the local site (see below)
7. procedure risk judged to be not high (see below)

Exclusion Criteria:

Patient exclusion criteria are:

Pre-catheterization

1. inability to give informed consent
2. ST-segment elevation myocardial infarction
3. pregnancy Post-catheterization
4. high likelihood of requiring a device not available at the hospitals without SOS (see below)
5. no need for PCI
6. need for coronary artery bypass surgery
7. high procedural risk (see below)

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population includes inpatients and outpatients undergoing diagnostic cardiac catheterization for suspected coronary artery disease (CAD) at hospitals without SOS.
Sampling Method: Non-Probability Sample
Enrollment: 31390 (Actual)
Dates: Start 2011-04-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Thru Index or Transfer Hospital Discharge on average 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Aversano, MD, Principal Investigator — Johns Hopkins University
Locations (37):
- United States (37):
  - Crestwood Medical Center, Huntsville, Alabama
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Hopkins Bayview Medical Center, Baltimore, Maryland
  - St. Agnes Hospital, Catonsville, Maryland
  - Southern Maryland Hospital Center, Clinton, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Baltimore Washington Medical Center, Glen Burnie, Maryland
  - Meritus Medical Center, Hagerstown, Maryland
  - Shady Grove Adventist Hospital, Rockville, Maryland
  - Bayonne Medical Center, Bayonne, New Jersey
  - Clara Maas Medical Center, Belleville, New Jersey
  - JFK Medical Center, Edison, New Jersey
  - Trinitas Hospital, Elizabeth, New Jersey
  - Virtua West Jersey Hospital, Marlton, New Jersey
  - Raritan Bay Medical Center, Perth Amboy, New Jersey
  - Riverview Medical Center, Red Bank, New Jersey
  - Somerset Medical Center, Somerville, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Holy Name Hospital, Teaneck, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Community Health and Wellness Center, Bryan, Ohio
  - University Hospital Geauga Medical Center, Chardon, Ohio
  - Ohio State University Hospital East, Columbus, Ohio
  - Mt. Carmel St. Ann Hospital, Columbus, Ohio
  - Southview Medical Center, Dayton, Ohio
  - Fort Hamilton Hospital, Hamilton, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - West Chester Hospital, West Chester, Ohio
  - Armstrong County Memorial Hospital, Kittanning, Pennsylvania
  - Evangelical Community Hospital, Lewisburg, Pennsylvania
  - UPMC McKeesport, McKeesport, Pennsylvania
  - Meadville Medical Center, Meadville, Pennsylvania
  - Monongahela Valley Hospital, Monongahela, Pennsylvania
  - Nazareth Hospital, Philadelphia, Pennsylvania
  - Memorial Hospital, York, Pennsylvania